CLINICAL TRIAL: NCT02683434
Title: Effects of Kinesio Taping on Postural Stability in Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Assistant Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA15/386
Record Dates: First submitted 2016-01-29; First posted 2016-02-17 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Increasing Performance of Healthy Athlete
Keywords: soccer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KT (Experimental): Kinesio Taping Application
  Interventions: Device: Kinesio Taping application
- CONTROL (No Intervention)

INTERVENTIONS:
Device: Kinesio Taping application — Therapeutic taping application applied to skin affecting muscle, fascia, circulation, ligaments, tendons and joints.
  Other Names: Kinesio Tex Gold, Kinesio Tex FP
  Arms: KT

SUMMARY:
The purpose of our study is to investigate the effects of Kinesio Taping application, which is applied before the training period, on postural stability in young soccer players.

ELIGIBILITY:
Inclusion Criteria:

- Soccer players aged between 12-16

Exclusion Criteria:

- Players who had lower extremity injury previously

Ages: 12 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Tetrax interactive balance system results | 45 minutes
  Postural Stability of soccer players

SECONDARY OUTCOMES:
Change in Flir E5 Thermographic Camera results | 45 minutes
  Skin temperature measurement of soccer players

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided